CLINICAL TRIAL: NCT06715371
Title: Reassessing Normative Cardiac Chamber Measurements: A Comparative Study of TTE and TEE Under General Anesthesia.
Brief Title: Comparing Cardiac Chamber Measurements: TTE vs. TEE Under Anesthesia
Acronym: CM-TTE-TEE
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 6347
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-11

CONDITIONS: Heart Chambers
Keywords: Cardiac Imaging; Cardiac Chamber Dimensions; General Anesthesia; Cardiac Surgery; Imaging Agreement; Diagnostic Accuracy; Perioperative Care; Echocardiography
MeSH Terms: interventions — Echocardiography; Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Surgery Patients: Patients undergoing cardiac surgery (eg., coronary revascularization) at Sunnybrook Health Sciences Centre.
  Interventions: Diagnostic Test: Transthoracic Echocardiography (TTE) and Transesophageal Echocardiography (TEE)

INTERVENTIONS:
Diagnostic Test: Transthoracic Echocardiography (TTE) and Transesophageal Echocardiography (TEE) — Transthoracic echocardiography (TTE) is a non-invasive imaging technique performed by placing an ultrasound transducer on the chest to obtain detailed heart images. TTE is conducted preoperatively on awake patients within two weeks prior to cardiac surgery, following ASE chamber quantification guidelines.
  Transesophageal echocardiography (TEE) is an invasive imaging technique where an ultrasound transducer is placed in the esophagus, providing closer and clearer images of the heart. TEE is performed intraoperatively under general anesthesia as part of routine care.
  Other Names: Transthoracic Echocardiography (TTE); Transesophageal Echocardiography (TEE)

SUMMARY:
This study aims to compare two common ultrasound techniques used during heart surgery: transthoracic echocardiography (TTE) and transesophageal echocardiography (TEE). TTE is performed by placing an ultrasound probe on the chest, while TEE involves inserting a probe into the esophagus, which provides closer and clearer images of the heart. Both methods are part of routine care for patients undergoing heart surgery.

The goal of this study is to assess how well the measurements from TTE and TEE agree in evaluating heart chamber dimensions during surgery and to investigate how factors such as anesthesia, breathing techniques affect these measurements.

This research involves 114 adult patients scheduled for heart surgery at Sunnybrook Health Sciences Centre. Participants will have TTE performed before and after surgery, and TEE will be conducted during surgery. All procedures are part of the usual standard of care.

By comparing these imaging techniques, the study seeks to provide more accurate and up-to-date guidelines for cardiac measurements, ensuring better care for patients during heart surgery.

DETAILED DESCRIPTION:
This observational study compares transthoracic echocardiography (TTE) and transesophageal echocardiography (TEE) in measuring cardiac chamber dimensions in adult patients undergoing cardiac surgery. While both techniques are integral to clinical care, TEE is typically used intraoperatively for its superior image quality, and TTE is performed preoperatively as a non-invasive diagnostic tool. However, differences in measurement values between TTE and TEE, particularly under the physiological changes induced by general anesthesia and positive end-expiratory pressure (PEEP), remain poorly understood. This study seeks to address this gap and update normative cardiac measurement values.

Study Design: A prospective observational study enrolling patients scheduled for coronary revascularization surgery at Sunnybrook Health Sciences Centre (n=114). All imaging procedures are part of routine clinical care.

Primary Objective: To evaluate the agreement between preoperative TTE and intraoperative TEE measurements of cardiac chamber dimensions.

Secondary Objectives:

* To explore how physiological changes from general anesthesia and PEEP impact the correlation between TTE and TEE measurements.
* To analyze how pre-existing cardiac conditions (e.g., hypertension, diabetes, atrial fibrillation) affect the agreement between these modalities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, able to provide informed consent.
* Patients scheduled for coronary revascularization cardiac surgery under general anesthesia.
* With normal left ventricular (LV) systolic function, defined by an ejection fraction of 50% or more, and normal right ventricular (RV) systolic function.
* Requiring intraoperative echocardiographic assessment.

Exclusion Criteria:

* Patients with contraindications to either transthoracic echocardiography (TTE) or transesophageal echocardiography (TEE).
* History of poor-quality echocardiography data that preclude accurate assessment.
* Undergoing emergency cardiac surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective cardiac surgery, specifically coronary revascularization procedures.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between preoperative TTE and intraoperative TEE measurements | Within 2 weeks prior to surgery and during surgery
  The correlation between preoperative transthoracic echocardiography (TTE) and intraoperative transesophageal echocardiography (TEE) measurements of cardiac chamber dimensions, including left ventricular internal dimensions, left atrial volume, and right atrial dimensions.

SECONDARY OUTCOMES:
Impact of general anesthesia on correlation between TTE and TEE. | Within 2 weeks prior to surgery and during surgery
  Impact of physiological changes induced by general anesthesia on the correlation between TTE and TEE measurements.
Impact of PEEP on correlation between TTE and TEE | Within 2 weeks prior to surgery and during surgery
  Impact of physiological changes induced by PEEP on the correlation between TTE and TEE measurements.
Impact of cardiac conditions on correlation between TTE and TEE. | Within 2 weeks prior to surgery and during surgery
  Impact of cardiac conditions (e.g., COPD, hypertension, history of atrial fibrillation) on the correlation between TTE and TEE measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo Moreno Garijo, MD, PhD, Principal Investigator — Sunnybrook Health Science Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data will be made available upon reasonable request to study PI following publication of full trial results.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available following publication of the full trial results.
Access Criteria: Data and supporting information will be made available following reasonable request directly to study PI.

REFERENCES:
- [Background] Kabirdas D, Scridon C, Brenes JC, Hernandez AV, Novaro GM, Asher CR. Accuracy of transthoracic echocardiography for the measurement of the ascending aorta: comparison with transesophageal echocardiography. Clin Cardiol. 2010 Aug;33(8):502-7. doi: 10.1002/clc.20807. PMID 20734448
- [Background] Singh H, Jain AC, Bhumbla DK, Failinger C. Comparison of left atrial dimensions by transesophageal and transthoracic echocardiography. Echocardiography. 2005 Nov;22(10):789-96. doi: 10.1111/j.1540-8175.2005.00128.x. PMID 16343160
- [Background] Shiran A, Adawi S, Ganaeem M, Asmer E. Accuracy and reproducibility of left ventricular outflow tract diameter measurement using transthoracic when compared with transesophageal echocardiography in systole and diastole. Eur J Echocardiogr. 2009 Mar;10(2):319-24. doi: 10.1093/ejechocard/jen254. Epub 2008 Oct 2. PMID 18835821
- [Background] Block M, Hourigan L, Bellows WH, Reeves J 3rd, Romson JL, Tran M, Pastor D, Schiller NB, Leung JM. Comparison of left atrial dimensions by transesophageal and transthoracic echocardiography. J Am Soc Echocardiogr. 2002 Feb;15(2):143-9. doi: 10.1067/mje.2002.121399. PMID 11836489
- [Background] Assanangkornchai N, Villeneuve V, McDonald S, Magder S, Shum Tim D, Buithieu J, Hatzakorzian R. Interchangeability of transthoracic and transesophageal echocardiographic right heart measurements in the perioperative setting and correlation with hemodynamic parameters. Int J Cardiovasc Imaging. 2023 Mar;39(3):555-563. doi: 10.1007/s10554-022-02754-1. Epub 2022 Nov 18. PMID 36399180
- [Background] Skarvan K, Lambert A, Filipovic M, Seeberger M. Reference values for left ventricular function in subjects under general anaesthesia and controlled ventilation assessed by two-dimensional transoesophageal echocardiography. Eur J Anaesthesiol. 2001 Nov;18(11):713-22. doi: 10.1046/j.1365-2346.2001.00915.x. PMID 11580777
- [Background] Cohen GI, White M, Sochowski RA, Klein AL, Bridge PD, Stewart WJ, Chan KL. Reference values for normal adult transesophageal echocardiographic measurements. J Am Soc Echocardiogr. 1995 May-Jun;8(3):221-30. doi: 10.1016/s0894-7317(05)80031-8. PMID 7640014
- [Background] Teran F, Prats MI, Nelson BP, Kessler R, Blaivas M, Peberdy MA, Shillcutt SK, Arntfield RT, Bahner D. Focused Transesophageal Echocardiography During Cardiac Arrest Resuscitation: JACC Review Topic of the Week. J Am Coll Cardiol. 2020 Aug 11;76(6):745-754. doi: 10.1016/j.jacc.2020.05.074. PMID 32762909
- [Background] Giron-Arango L, D'Empaire PP. Is There a Role for Transesophageal Echocardiography in the Perioperative Trauma Patient? Curr Anesthesiol Rep. 2022;12(2):210-216. doi: 10.1007/s40140-022-00526-0. Epub 2022 Mar 19. PMID 35340714

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT06715371/Prot_SAP_000.pdf